CLINICAL TRIAL: NCT04341441
Title: Will Hydroxychloroquine Impede or Prevent COVID-19: WHIP COVID-19 Study
Brief Title: Will Hydroxychloroquine Impede or Prevent COVID-19
Acronym: WHIP COVID-19
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis did not reveal any safety concerns by the DSMB, but unblinded data did not provide support to continue. Event rate did not meet projected magnitude; given low recruitment potential, it is unlikely that a positive result will occur.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, William W. O'Neill, Director, Center for Structural Heart Disease, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1410401
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: COVID-19; Coronavirus; Coronavirus Infections; SARS-CoV 2
Keywords: COVID-19; Coronavirus; Healthcare Workers; SARS-CoV 2; First Responders; Emergency Medical Technicians; Paramedics; Firefighters; Police Officers; Detroit; Michigan; Henry Ford Hospital
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: This is a prospective, multi-site study designed to evaluate whether the use of hydroxychloroquine in healthcare workers (HCW) and first responders (FR) in southeast (SE) Michigan, can prevent the acquisition, symptoms and clinical COVID-19 infection.
  The study will randomize a total of 3,000 Healthcare Workers and First Responders, age ≥18 years or older, through the Henry Ford Health System, Detroit COVID Consortium. The participants who meeting study entry criteria and are not on HCQ prior to study enrollment will be randomized in a 1:1:1 blinded comparison of daily or weekly oral hydroxychloroquine versus oral placebo for 8 weeks.
  A fourth non-randomized comparator group will be enrolled in the study comprising of HCW who are chronically on HCQ as part of their standard of care for their autoimmune disease(s). This will be an open enrollment group and will provide information of chronic weight-based daily therapy of HCQ effectiveness as a prophylactic/preventive strategy.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinded randomization will be performed by the Henry Ford Hospital Public Health Sciences investigators once the participants are determined to be eligible for enrollment. Randomization will be stratified by study site and risk of exposure based on location of work and type of work.
  Once enrolled, each Participant will be assigned a unique identifier (detailed in the full protocol). This number, along with the assigned site number, will constitute the Subject Identifier (Subject ID).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Study Drug - Daily Dose (Active Comparator): The daily hydroxychloroquine treatment arm will receive a 200 mg oral dose daily following day 1 dose of 400 mg orally once. This dose represents approximately half the standard weight-based dosing recommended for management of autoimmune diseases and therefore less likely to produce side effects than standard of care.
  Interventions: Drug: Hydroxychloroquine - Daily Dosing; Diagnostic Test: Monitoring Visit - Baseline; Diagnostic Test: Monitoring Visit - Week 4; Diagnostic Test: Monitoring Visit - Week 8; Other: Weekly Assessment
- Study Drug - Weekly Dose (Active Comparator): The once weekly randomized treatment arm will receive the proposed dose of hydroxychloroquine for prophylaxis of malaria is 6.5 mg/kg per dose (maximum of 400mg per dose) administered orally weekly on the same day of each week. This is based on the recommended dose for prophylaxis of malaria.
  Interventions: Drug: Hydroxychloroquine - Weekly Dosing; Diagnostic Test: Monitoring Visit - Baseline; Diagnostic Test: Monitoring Visit - Week 4; Diagnostic Test: Monitoring Visit - Week 8; Other: Weekly Assessment
- Placebo (Active Comparator): All treatment groups will receive placebo pills to have the patients take 2 pills a day. The randomized placebo arm will receive placebo pills made to resemble the daily dosing of HCQ. Similarly, the once a week treatment arm will receive placebo pills for the days not on HCQ medication.
  Interventions: Other: Placebo oral tablet; Diagnostic Test: Monitoring Visit - Baseline; Diagnostic Test: Monitoring Visit - Week 4; Diagnostic Test: Monitoring Visit - Week 8; Other: Weekly Assessment
- Non-Randomized Active Comparator (Active Comparator): A non-randomized comparator group will be enrolled in the study comprising of healthcare workers and first responders who are chronically on oral hydroxychloroquine as part of their standard of care for their autoimmune disease(s). This will be an open enrollment group and will provide information of chronic weight-based daily therapy of HCQ effectiveness as a prophylactic/preventive strategy.
  Interventions: Diagnostic Test: Monitoring Visit - Baseline; Diagnostic Test: Monitoring Visit - Week 4; Diagnostic Test: Monitoring Visit - Week 8; Other: Weekly Assessment

INTERVENTIONS:
Drug: Hydroxychloroquine - Daily Dosing — The daily hydroxychloroquine treatment arm will receive a 200 mg oral dose daily following day 1 dose of 400 mg orally once. This dose represents approximately half the standard weight-based dosing recommended for management of autoimmune diseases and therefore less likely to produce side effects than standard of care.
  All treatment groups will receive placebo pills to have the patients take 2 pills a day.
  Other Names: Study Drug - Daily; Daily Oral Dosing
  Arms: Study Drug - Daily Dose
Drug: Hydroxychloroquine - Weekly Dosing — The once weekly randomized treatment arm will receive the proposed dose of hydroxychloroquine for prophylaxis of malaria is 6.5 mg/kg per dose (maximum of 400 mg per dose) administered orally weekly on the same day of each week. This is based on the recommended dose for prophylaxis of malaria
  All treatment groups will receive placebo pills to have the patients take 2 pills a day.
  Other Names: Weekly Oral Dosing
  Arms: Study Drug - Weekly Dose
Other: Placebo oral tablet — Participants randomized to this arm will be provided with daily dosing of oral placebo to have the patients take 2 pills a day..
  Participants will receive a monitoring phone call at 4 weeks post study entry to monitor for COVID-19 symptoms and medication side effects. At week 8, participants will provide additional samples of whole blood.
  Additional studies will include serology, inflammatory and other disease associated markers. Clinical data and location of main work area will be collected.
  Other Names: Placebo
  Arms: Placebo
Diagnostic Test: Monitoring Visit - Baseline — Face-to-face monitoring visit to obtain monitoring questionnaires to assess for COVID-19 symptoms/diagnosis, adherence and medication side effects, and collect study blood samples. Three (3) blood specimens will be collected from each Participant using the sterile procedure as routine standard of care. A total of five (5) 10 mL tubes of whole blood will be collected at each timepoint.
  Other Names: Baseline Monitoring Visit
Diagnostic Test: Monitoring Visit - Week 4 — Face-to-face monitoring visit to obtain monitoring questionnaires to assess for COVID-19 symptoms/diagnosis, adherence and medication side effects, and collect study blood samples. Three (3) blood specimens will be collected from each Participant using the sterile procedure as routine standard of care. A total of five (5) 10 mL tubes of whole blood will be collected at each timepoint.
  Other Names: Week 4 - Monitoring Visit
Diagnostic Test: Monitoring Visit - Week 8 — Face-to-face monitoring visit to obtain monitoring questionnaires to assess for COVID-19 symptoms/diagnosis, adherence and medication side effects, and collect study blood samples. Three (3) blood specimens will be collected from each Participant using the sterile procedure as routine standard of care. A total of five (5) 10 mL tubes of whole blood will be collected at each timepoint.
  Other Names: Week 8 - Monitoring Visit
Other: Weekly Assessment — Participants will be asked to contact the study team if COVID-19 infection is established at any time during the study. For study weeks 1,2,3,5,6 &7, Participants will receive a monitoring questionnaire to assess for COVID-19 symptoms/diagnosis, adherence and medication side effects. These monitoring visits will be done by telephone and/or electronic encounters (virtual visits, email), whichever method the patient prefers to encourage adherence to the monitoring.
  Other Names: Monitoring Call

SUMMARY:
This is a prospective, multi-site study designed to evaluate whether the use of hydroxychloroquine in healthcare workers (HCW), Nursing Home Workers (NHW), first responders (FR), and Detroit Department of Transportation bus drivers (DDOT) in SE, Michigan, can prevent the acquisition, symptoms and clinical COVID-19 infection

The primary objective of this study is to determine whether the use of daily or weekly oral hydroxychloroquine (HCQ) therapy will prevent SARS-CoV-2 infection and COVID-19 viremia and clinical COVID-19 infection healthcare workers (HCW) and first responders (FR) (EMS, Fire, Police, bus drivers) in Southeast Michigan.

Preventing COVID-19 transmission to HCW, FR, and Detroit Department of Transportation (DDOT) bus drivers is a critical step in preserving the health care and first responder force, the prevention of COVID-19 transmission in health care facilities, with the potential to preserve thousands of lives in addition to sustaining health care systems and civil services both nationally and globally. If efficacious, further studies on the use of hydroxychloroquine to prevent COVID-19 in the general population could be undertaken, with a potential impact on hundreds of thousands of lives.

DETAILED DESCRIPTION:
The study will randomize a total of 3,000 HCW, NHW, FR and DDOT bus drivers within Henry Ford Hospital System, the Detroit COVID Consortium in Southeast, Michigan. The participants will be randomized in a 1:1:1 blinded comparison of daily HCQ, weekly HCQ, or placebo. A fourth non-randomized comparator group of HCW, NHW, DDOT bus drivers, and FR who are currently on standard HCQ therapy will be recruited to assess the impact of weightbased daily dosing of HCQ as compared to the randomized arms.

Eligible participants who are asymptomatic for pre-specified signs and symptoms suggestive of COVID-19 infection will have a whole blood specimen obtained at study entry.

Participants will be provided with weekly dosing of hydroxychloroquine (HCQ) 400mg po q weekly, daily dosing of HCQ 200mg po q daily following a loading dose of 400mg day 1, or placebo. Participants will receive monitoring at each study week visit to assess for the development of COVID-19 related symptoms, COVID-19 clinical disease, and medication side effects. At week 8 or if diagnosed positive, participants will provide additional samples of whole blood and complete the final study questionnaire.

Data including demographic, clinical results, work duties, location of main work area and possible exposures in the community will be collected through questionnaires and EMR review. Disease-specific, immunologic, and other serologic marker data will be obtained from stored samples.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to provide informed consent.
2. Participant is 18-75 years of age.
3. Participant does not have symptoms of respiratory infection, including cough, fevers (temperature >38.0C), difficulty breathing, shortness of breath, chest pains, malaise, myalgia, headaches, nausea or vomiting, or other symptoms associated with COVID-19.
4. Participant is willing to provide blood samples for the study.
5. Subject agrees to all aspects of the study.
6. The participant has no known allergies or contraindications (as stated in the consent form) to the use of hydroxychloroquine (HCQ) as noted in the exclusion criteria and Pharmacy sections.

Exclusion Criteria:

1. Does not meet inclusion criteria.
2. Participant unable or unwilling to provide informed consent.
3. Participant has any of the symptoms above or screens positive for possible COVID-19 disease.
4. Participant is currently enrolled in a study to evaluate an investigational drug.
5. Vulnerable populations deemed inappropriate for study by the site Principal Investigator.
6. The participant has a known allergy/hypersensitivity or has a medication or co-morbidity (including history of gastric bypass, epilepsy, cardiovascular disease or renal failure) that prevents the use of HCQ (see pharmacy section).
7. The participant is a woman of childbearing age whose pregnancy status is unknown and is not willing to use 2 methods of contraception.
8. The participant is pregnant or nursing.
9. The participant was diagnosed with retinopathy prior to study entry.
10. The participant has a diagnosis of porphyria prior to study entry.
11. The participant has renal failure with a creatinine clearance of <10 ml/min, pre-dialysis or requiring dialysis.
12. The Participant has a family history of Sudden Cardiac Death.
13. The participant is currently on diuretic therapy.
14. The participant has a history of known Prolonged QT Syndrome.
15. The participant is already taking any of the following medications: Abiraterone acetate, Agalsidase, Amodiaquine, Azithromycin, Conivaptan, Dabrafenib, Dacomitinib, Dapsone (Systemic), Digoxin, Enzalutamide, Fusidic Acid (Systemic), Idelalisib, Lanthanum, Lumefantrine, Mefloquine, Mifepristone, Mitotane, Pimozide, QT-prolonging Agents, Stiripentol).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William W O'Neill, MD, Principal Investigator — Henry Ford Health System; Dee Dee Wang, MD, Study Director — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bai Y, Yao L, Wei T, Tian F, Jin DY, Chen L, Wang M. Presumed Asymptomatic Carrier Transmission of COVID-19. JAMA. 2020 Apr 14;323(14):1406-1407. doi: 10.1001/jama.2020.2565. PMID 32083643
- [Background] Chang D, Xu H, Rebaza A, Sharma L, Dela Cruz CS. Protecting health-care workers from subclinical coronavirus infection. Lancet Respir Med. 2020 Mar;8(3):e13. doi: 10.1016/S2213-2600(20)30066-7. Epub 2020 Feb 13. No abstract available. PMID 32061333
- [Background] Liu J, Cao R, Xu M, Wang X, Zhang H, Hu H, Li Y, Hu Z, Zhong W, Wang M. Hydroxychloroquine, a less toxic derivative of chloroquine, is effective in inhibiting SARS-CoV-2 infection in vitro. Cell Discov. 2020 Mar 18;6:16. doi: 10.1038/s41421-020-0156-0. eCollection 2020. No abstract available. PMID 32194981
- [Background] Vincent MJ, Bergeron E, Benjannet S, Erickson BR, Rollin PE, Ksiazek TG, Seidah NG, Nichol ST. Chloroquine is a potent inhibitor of SARS coronavirus infection and spread. Virol J. 2005 Aug 22;2:69. doi: 10.1186/1743-422X-2-69. PMID 16115318
- [Background] Ben-Zvi I, Kivity S, Langevitz P, Shoenfeld Y. Hydroxychloroquine: from malaria to autoimmunity. Clin Rev Allergy Immunol. 2012 Apr;42(2):145-53. doi: 10.1007/s12016-010-8243-x. PMID 21221847
- [Background] Mohammad S, Clowse MEB, Eudy AM, Criscione-Schreiber LG. Examination of Hydroxychloroquine Use and Hemolytic Anemia in G6PDH-Deficient Patients. Arthritis Care Res (Hoboken). 2018 Mar;70(3):481-485. doi: 10.1002/acr.23296. Epub 2018 Feb 9. PMID 28556555
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618
- [Background] Lim HS, Im JS, Cho JY, Bae KS, Klein TA, Yeom JS, Kim TS, Choi JS, Jang IJ, Park JW. Pharmacokinetics of hydroxychloroquine and its clinical implications in chemoprophylaxis against malaria caused by Plasmodium vivax. Antimicrob Agents Chemother. 2009 Apr;53(4):1468-75. doi: 10.1128/AAC.00339-08. Epub 2009 Feb 2. PMID 19188392
- [Background] Howard DR, Brown JM, Todd S, Gregory WM. Recommendations on multiple testing adjustment in multi-arm trials with a shared control group. Stat Methods Med Res. 2018 May;27(5):1513-1530. doi: 10.1177/0962280216664759. Epub 2016 Sep 19. PMID 27647808

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Drug - Daily Dose: 200 mg oral dose daily following day 1 dose of 400 mg orally once. This dose represents approximately half the standard weight-based dosing recommended for management of autoimmune diseases and therefore less likely to produce side effects than standard of care.
  All treatment groups will receive placebo pills to have the patients take 2 pills a day.
- Study Drug - Weekly Dose: 6.5 mg/kg per dose (maximum of 400mg per dose) administered orally weekly on the same day of each week. This is based on the recommended dose for prophylaxis of malaria.
  All treatment groups will receive placebo pills to have the patients take 2 pills a day.
- Placebo: Placebo oral tablet: Participants randomized to this arm will be provided with daily dosing of oral placebo to have the patients take 2 pills a day.
  All treatment groups will receive placebo pills to have the patients take 2 pills a day. The randomized placebo arm will receive placebo pills made to resemble the daily dosing of HCQ. Similarly, the once a week treatment arm will receive placebo pills for the days not on HCQ medication.
- Non-Randomized Active Comparator (HCQ Cohort): This non-randomized comparator group is comprised of healthcare workers and first responders who are chronically on oral hydroxychloroquine as part of standard of care for autoimmune disease(s).
Period: Overall Study
Arm/Group | Study Drug - Daily Dose | Study Drug - Weekly Dose | Placebo | Non-Randomized Active Comparator (HCQ Cohort)
Started | 197 | 201 | 200 | 26
Completed | 188 | 199 | 191 | 26
Not Completed | 9 | 2 | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-Randomized Active Comparator: This will be an open enrollment group and will provide information of chronic weight-based daily therapy of HCQ effectiveness as a prophylactic/preventive strategy.
  This non-randomized comparator group will be enrolled in the study comprising of healthcare workers and first responders who are chronically on oral hydroxychloroquine as part of their standard of care for their autoimmune disease(s).
- Total: Total of all reporting groups
Arm/Group | Study Drug - Daily Dose | Study Drug - Weekly Dose | Placebo | Non-Randomized Active Comparator | Total
Number analyzed (Participants) | 197 | 201 | 200 | 26 | 624
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (11.5) | 45.7 (11.7) | 43.7 (12.7) | 45.8 (11.7) | 44.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 110 | 120 | 23 | 370
  Male | 80 | 91 | 80 | 3 | 254
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 11 | 5 | 10 | 6 | 32
  White | 163 | 179 | 169 | 18 | 529
  AS/IN/PI | 15 | 10 | 15 | 2 | 42
Region of Enrollment [Number; unit: participants]
  United States | 197 | 201 | 200 | 26 | 624

OUTCOME MEASURES:

1. Primary Outcome: To Determine if the Use of Hydroxychloroquine as Preventive Therapy Decreases the Rate of Acquisition of SARS-CoV 2 Infections With Clinical COVID-19 Disease in Study Participants for Each Randomized Treatment Arm as Compared to Placebo.
Description: The rate of acquisition of SARS-CoV 2 infections and clinical COVID-19 disease (number of events) in study participants for each randomized hydroxychloroquine treatment arm was compared to the placebo treatment arm. This included both symptomatic and asymptomatic patients.
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug - Daily Dose | Study Drug - Weekly Dose | Placebo | Non-Randomized Active Comparator
Number analyzed (Participants) | 188 | 199 | 191 | 25
Participants | 1 | 1 | 1 | 0
Statistical Analysis 1: Comparison: Study Drug - Daily Dose vs Study Drug - Weekly Dose vs Placebo vs Non-Randomized Active Comparator; Test type: Superiority — Sample size was determined with one planned interim analysis when 50% of participants had completed their 8 weeks of treatment using an O'Brien-Fleming alpha spending method to ensure an overall type 1 error of 0.05. With a sample size of 900 per group and alpha = 0.0492, the power to detect a 32% reduction in COVID-19 disease rate (10% vs 6.8%) between the placebo and HCQ treated groups, determined at 87%. Study required 1000 per group with a total of 3000 patients to complete the trial; p = 0.75, Mantel Haenszel — P-value for the comparison between groups, including the non-randomized active comparator, was 0.75; Risk Ratio (RR) = 0.32 — Low number of primary events precluded estimated value of risk ratio

2. Secondary Outcome: Determine the Effect of Hydroxychloroquine Dose in the Prevention of COVID-19 Viremia and Disease.
Description: Compare the rates of SARS-CoV 2 symptomatic infections (number of events with both symptoms and positive test for COVID-19) between the randomized hydroxychloroquine treatment arms and the placebo control arm to determine the effect of HCQ dose in the prevention of COVID-19 viremia and disease. This analysis only includes only the randomized arms in the study (Study Drug - Daily Dose, Study Drug - Weekly Dose, and Placebo).
Time Frame: 8 Weeks
Population: Compare the rates of SARS-CoV 2 symptomatic infections (number of events with both symptoms and positive test for COVID-19) between the randomized hydroxychloroquine treatment arms and the placebo control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug - Daily Dose | Study Drug - Weekly Dose | Placebo
Number analyzed (Participants) | 188 | 199 | 191
Participants | 1 | 1 | 1

3. Secondary Outcome: Assess the Impact of Chronic Weight-based Dosing of HCQ for COVID-19 Prevention.
Description: Compare the rates of SARS-CoV 2 infections (number of events of symptomatic patients with a positive COVID-19 test) in the non-randomized comparator arm to the randomized hydroxychloroquine and placebo arms to assess the impact of chronic weight-based dosing of HCQ for COVID-19 prevention via weekly questionnaire and/or blood samples. This analysis includes all randomized and non-randomized groups in the study.
Time Frame: 8 Weeks
Population: This analysis outcome measure reports the number of occurrences of symptomatic patients with a positive COVID-19 test in all randomized and non-randomized groups in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug - Daily Dose | Study Drug - Weekly Dose | Placebo | Non-Randomized Active Comparator
Number analyzed (Participants) | 188 | 199 | 191 | 25
Participants | 1 | 1 | 1 | 0

4. Secondary Outcome: Comparison of the Rate of SARS-CoV 2 Infections as Measured by IgM/IgG Seroconversion in Study Participants Receiving Randomized HCQ Versus Placebo.
Description: Measurement of the rate of SARS-CoV 2 infections as measured by IgM/IgG seroconversion in study participants receiving randomized HCQ versus placebo via blood samples in the randomized arms of the study (Study Drug - Daily Dose, Study Drug - Weekly Dose, and Placebo).
Time Frame: 8 Weeks
Population: This analysis is only for the randomized arms of the study (Study Drug - Daily Dose, Study Drug - Weekly Dose, and Placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug - Daily Dose | Study Drug - Weekly Dose | Placebo
Number analyzed (Participants) | 188 | 199 | 191
Participants | 1 | 1 | 2

5. Secondary Outcome: Compare the Seroprevalence of SARS-CoV 2 IgM and/or IgG Positive Samples at Study Entry and Study Conclusion in All Participants Receiving HCQ Compared to Those Receiving Placebo.
Description: Measurement of the seroprevalence of SARS-CoV 2 IgM and/or IgG positive samples in all arms of the study, randomized and non-randomized (Study Drug - Daily Dose, Study Drug - Weekly Dose, Placebo, and Non-Randomized Active Comparator).
Time Frame: 8 Weeks
Population: The analysis reports the number of patient samples that seroconverted to positive serology for IgM and/or IgG by the subject end of study time point in all arms of the study, randomized and non-randomized (Study Drug - Daily Dose, Study Drug - Weekly Dose, Placebo, and Non-Randomized Active Comparator).
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug - Daily Dose | Study Drug - Weekly Dose | Placebo | Non-Randomized Active Comparator
Number analyzed (Participants) | 188 | 199 | 191 | 25
Participants | 1 | 1 | 2 | 0

6. Secondary Outcome: Comparison of the Emergence of Clinical Symptoms or COVID-19 Diagnosis in Participants Presenting Asymptomatically at Study Entry But Identified as Seropositive by Serology at Entry Between the Randomized Treatment Arms and Comparator Arm.
Description: Measurement of the emergence of clinical symptoms or COVID-19 diagnosis in participants presenting asymptomatically at study entry but identified as seropositive by serology at entry between the randomized treatment arms and comparator arm and via weekly questionnaire and/or blood samples.
Time Frame: 8 Weeks
Population: All patients were asymptomatic at study entry by observed lack of symptoms and consistent with study eligibility criteria. This analysis planned to evaluate patients who tested positive for COVID-19 at study entry time point, but had yet to develop symptoms when entering the study to assess efficacy of hydroxychloroquine in preventing symptom emergence. Only one participant met the criteria for outcome measure analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug - Daily Dose | Study Drug - Weekly Dose | Placebo | Non-Randomized Active Comparator
Number analyzed (Participants) | 188 | 199 | 191 | 25
Participants | 1 | 0 | 0 | 0

7. Secondary Outcome: To Examine the Level of Care Needed by Participants in Each Arm Developing COVID19 as Measured as Requiring Emergency Room Visit, Hospitalization or Able to Stay Home Without Hospital Care.
Description: Review of the level of care needed by participants in each arm developing COVID19 as measured as requiring emergency room visit, hospitalization or able to stay home without hospital care via weekly questionnaire.
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug - Daily Dose | Study Drug - Weekly Dose | Placebo | Non-Randomized Active Comparator
Number analyzed (Participants) | 188 | 199 | 191 | 25
Participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Determine the Safety and Tolerability of HCQ Dosing for Preventive Strategy Against COVID-19 as Measured by Adverse Events and Serious Adverse Events.
Description: Measurement of the safety and tolerability of HCQ dosing for preventive strategy against COVID-19 as measured by adverse events and serious adverse events reported via weekly questionnaire.
Time Frame: 8 Weeks
Measure: Number; unit: Number of adverse events.
Arm/Group | Study Drug - Daily Dose | Study Drug - Weekly Dose | Placebo | Non-Randomized Active Comparator
Number analyzed (Participants) | 188 | 199 | 191 | 26
Number of adverse events.
  Adverse events (only Level 1 and 2) observed in the study. | 206 | 193 | 188 | 2
  Serious adverse events (Level 3 or 4). | 0 | 0 | 0 | 0

9. Secondary Outcome: To Examine Other Clinical Factors Contributing to the Risk of SARS-CoV 2 Infection in Healthcare Workers and First Responders.
Description: Examination of other clinical factors contributing to the risk of SARS-CoV 2 infection including demographics, work type and location, positive COVID-19 partners, possible exposures and clinical symptoms via study visits and weekly questionnaire.
Time Frame: 8 Weeks
Population: Due to low number of events, this analysis was not performed. No factors were identified.
Measure: Number; unit: Clinical factors
Arm/Group | Study Drug - Daily Dose | Study Drug - Weekly Dose | Placebo | Non-Randomized Active Comparator
Number analyzed (Participants) | 188 | 199 | 191 | 25
Clinical factors | NA — Due to low number of events, this analysis was not performed. No factors were identified. | NA — Due to low number of events, this analysis was not performed. No factors were identified. | NA — Due to low number of events, this analysis was not performed. No factors were identified. | NA — Due to low number of events, this analysis was not performed. No factors were identified.

10. Secondary Outcome: Examine the Correlation Between HCQ Drug Levels and Development of COVID-19 Symptoms or Positive COVID-19 Test Results.
Description: Examination of the correlation between HCQ drug levels and development of COVID-19 clinical symptoms and/or positive COVID-19 test results via weekly subject questionnaire and/or blood samples.
Time Frame: 8 Weeks
Population: This analysis was not performed due to low number of events and early termination of the study. Therefore, no data or measures to report.
Measure: Number; unit: Correlation coefficient
Arm/Group | Study Drug - Daily Dose | Study Drug - Weekly Dose | Placebo | Non-Randomized Active Comparator
Number analyzed (Participants) | 188 | 199 | 191 | 25
Correlation coefficient | NA — Due to low number of events, this analysis was not performed. | NA — Due to low number of events, this analysis was not performed. . | NA — Due to low number of events, this analysis was not performed. | NA — Due to low number of events, this analysis was not performed.

11. Secondary Outcome: Identify Immunologic, Serological and Inflammatory Markers Associated With Acquisition and Response to COVID-19 in Both HCQ and Placebo Participants Developing Laboratory or Clinical Confirmed Disease.
Description: Identification of immunologic, serological and inflammatory markers associated with acquisition and response to COVID-19 in both HCQ and placebo Participants developing laboratory or clinical confirmed disease via study visits, weekly questionnaire, and blood samples.
Time Frame: 8 weeks
Population: This analysis was not performed due to low number of events and early termination of the study. Therefore, no data or markers to report.
Measure: Number; unit: Inflammatory markers
Arm/Group | Study Drug - Daily Dose | Study Drug - Weekly Dose | Placebo | Non-Randomized Active Comparator
Number analyzed (Participants) | 188 | 199 | 191 | 25
Inflammatory markers | NA — This analysis was not performed due to low number of events and early termination of the study. | NA — This analysis was not performed due to low number of events and early termination of the study. | NA — This analysis was not performed due to low number of events and early termination of the study. | NA — This analysis was not performed due to low number of events and early termination of the study.

ADVERSE EVENTS:
Time Frame: 8 weeks.
Groups:
- Non-Randomized Active Comparator (HCQ Cohort): This non-randomized comparator group is comprised of healthcare workers and first responders who are chronically on oral hydroxychloroquine as part of their standard of care for autoimmune disease(s).
Arm/Group | Study Drug - Daily Dose | Study Drug - Weekly Dose | Placebo | Non-Randomized Active Comparator (HCQ Cohort)
All-Cause Mortality (participants affected / at risk) | 0/188 | 0/199 | 0/191 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/188 | 0/199 | 0/191 | 0/26
Other Adverse Events (participants affected / at risk) | 97/188 | 95/199 | 85/191 | 2/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Drug - Daily Dose (N=188) | Study Drug - Weekly Dose (N=199) | Placebo (N=191) | Non-Randomized Active Comparator (HCQ Cohort) (N=26)
All gastrointestinal symptoms reported (Gastrointestinal disorders) | 36 (54) | 34 (43) | 42 (52) | 0 (0)
All cardiac symptoms reported (Cardiac disorders) | 16 (17) | 15 (16) | 10 (10) | 0 (0)
All ear and labyrinth symptoms reported (Ear and labyrinth disorders) | 9 (10) | 6 (9) | 8 (8) | 0 (0)
All eye symptoms reported (Eye disorders) | 6 (9) | 1 (1) | 6 (6) | 0 (0)
All general symptoms and administration site symptoms reported (General disorders) | 8 (9) | 13 (15) | 15 (17) | 0 (0)
All immune system symptoms reported (Immune system disorders) | 4 (4) | 5 (6) | 0 (0) | 0 (0)
All infection and infestation symptoms reported (Infections and infestations) | 8 (8) | 1 (1) | 3 (3) | 0 (0)
Injury, poisoning and procedural complication symptoms reported (Injury, poisoning and procedural complications) | 3 (3) | 1 (2) | 1 (1) | 1 (1)
Metabolism and nutrition symptoms reported (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
All Musculoskeletal and connective tissue symptoms reported (Musculoskeletal and connective tissue disorders) | 11 (13) | 16 (17) | 14 (16) | 1 (1)
All nervous system symptoms reported (Nervous system disorders) | 41 (43) | 30 (33) | 34 (42) | 0 (0)
All psychiatric symptoms reported (Psychiatric disorders) | 5 (6) | 10 (13) | 7 (7) | 0 (0)
All reproductive system and breast symptoms reported (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
All respiratory, thoracic and mediastinal symptoms reported (Respiratory, thoracic and mediastinal disorders) | 13 (17) | 22 (27) | 15 (21) | 0 (0)
All skin and subcutaneous tissue symptoms reported (Skin and subcutaneous tissue disorders) | 11 (12) | 7 (10) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Study has been terminated. Interim analysis did not reveal any safety concerns by the DSMB with hydroxychloroquine treatment, but unblinded data did not provide support to continue due to low numbers of events. Event rate did not meet projected magnitude; given low recruitment potential, it is unlikely that a positive result will occur.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT04341441/Prot_001.pdf
  • Statistical Analysis Plan (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT04341441/SAP_002.pdf